CLINICAL TRIAL: NCT03907540
Title: Open-label, 2-part Study Designated to Assess the Absolute Bioavailability of KD025 and to Determine the Mass Balance Recovery, Metabolite Profile and Identification of Metabolite Structures for [14C]-KD025 in Healthy Male Subjects
Brief Title: Human Absorption, Distribution and Metabolism Study (hAME) [14C]-KD025
Acronym: KD025-108
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: KD025-108; 2018-004773-28 (EudraCT Number)
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Autoimmune Diseases; Fibrosis
Keywords: absorption; metabolism; excretion
MeSH Terms: conditions — Autoimmune Diseases; Fibrosis | interventions — belumosudil; Tablets; KD025

STUDY DESIGN:
Intervention Model Description: Single center, non-randomized, open-label, 2-part study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1, Treatment A--Belumosudil 200 mg Tablet (Experimental): Belumosudil 200 mg tablet
  Interventions: Drug: Belumosudil 200 mg tablet
- Part 1, Treatment B--[14C]-KD025 IV Microdose (Experimental): [14C]-KD025 at a dose of 100 μg in a 5 mL solution containing NMT 37 kBq (1000 nCi) [14C] over 15 min IV
  Interventions: Drug: [14C]-KD025 at a dose of 100 μg in a 5 mL solution IV microdose
- Part 2, Treatment C--[14C]-KD025 Capsule (Experimental): [14C]-KD025 200 mg capsule containing NMT 9.8 MBq (215 μCi)
  Interventions: Drug: [14C]-KD025 200 mg capsule

INTERVENTIONS:
Drug: Belumosudil 200 mg tablet — Belumosudil 200 mg tablet, development candidate
  Other Names: Rezurock (brand name); KD025; SLx-2119
  Arms: Part 1, Treatment A--Belumosudil 200 mg Tablet
Drug: [14C]-KD025 at a dose of 100 μg in a 5 mL solution IV microdose — test investigational medicinal product
  Arms: Part 1, Treatment B--[14C]-KD025 IV Microdose
Drug: [14C]-KD025 200 mg capsule — test investigational medicinal product
  Arms: Part 2, Treatment C--[14C]-KD025 Capsule

SUMMARY:
Human, absorption, metabolism and excretion study of belumosudil (KD025)

DETAILED DESCRIPTION:
This is an open-label, 2-part study designed to assess the absolute bioavailability of belumosudil (KD025) and to determine the mass balance recovery, metabolite profile, and identification of metabolite structures for [14C]-KD025 in healthy male subjects.

Primary Objectives

* To determine the absolute oral bioavailability of KD025 (Part 1)
* To determine the mass balance recovery after a single oral dose of [14C]-KD025 (Part 2)
* To provide plasma, urine, and fecal samples for metabolite profiling and structural identification (Part 2)

Secondary Objectives

* To obtain information regarding the oral PK of total radioactivity, KD025 and its metabolites KD025m1 and KD025m2, in plasma
* To obtain information regarding the intravenous (IV) pharmacokinetics (PK) of [14C]-KD025 in plasma (Part 1)
* To determine the routes and rates of elimination of [14C]-KD025 and associated total radioactivity (Part 2)
* To evaluate the extent of distribution of total radioactivity into blood cells (Part 2)
* To assess the qualitative and quantitative metabolic profile of [14C]-KD025 and carry out the structural elucidation of the main metabolites in plasma (accounting for ≥ 10% of circulating total radioactivity) and in urine and fecal samples accounting for ≥ 10% of administered dose (Part 2)
* To provide additional safety and tolerability information for belumosudil

PART 1:

Part 1 is an open-label, non-randomized single oral dose followed by an IV microtracer assessment in 5 healthy male subjects. Subjects receive a single oral dose of belumosudil (KD025) 200 mg Tablet (Treatment A), in the fed state following a standard breakfast on the morning of Day 1. Subjects then receive an IV dose of 100 μg [14C]-KD025 (a 'microdose') containing not more than (NMT) 37 kBq (kilobecquerel; 1000 nanocurie [nCi]) [14C], as a 15 min IV infusion (Treatment B), beginning 1.75 hours (h) after the oral dose administration (Treatment A), i.e., 15 minutes [min] before the expected time of maximum concentration [Tmax] 2 h) for the oral dose.

Planned enrollment is to be 6 subjects to ensure 4 evaluable subjects. An evaluable subject for Part 1 will be defined as a subject who had sufficient data for evaluation of the primary oral bioavailability objective of the study.

All subjects are to undergo preliminary screening procedures to determine their eligibility for Part 1 and Part 2 at the screening visit (Day -28 to Day -2 of Part 1). Subjects are to be admitted to the clinical unit on the evening prior to investigational medicinal product (IMP) administration (Day -1 of Part 1) for confirmation of eligibility and baseline procedures. Subjects will be dosed on the morning following admission (Day 1 of Part 1). Following an overnight fast (approximately 10 h), subjects are to consume a standard breakfast and receive a single dose of Belumosudil 200 mg Tablet (Treatment A) 30 min after the start of breakfast. At 1 h 45 min (1.75 h) after Treatment A administration, subjects are to receive an IV infusion of [14C]-KD025 solution, 100 µg (Treatment B). Subjects are to remain resident in the clinic until up to 48 hours post-oral dose (up to Day 3). The minimum washout period between dose administrations in Part 1 and 2 is 7 days.

PART 2:

Part 2 is an open-label, non-randomized absorption, distribution, metabolism, and elimination (ADME) assessment in 5 healthy male subjects. Following a minimum washout period of 7 days, subjects who participated in Part 1 of the study are to be admitted to the clinical unit for participation in Part 2 of the study. Subjects are to receive a single oral administration of [14C]-KD025 200 mg Capsule containing NMT 9.8 MBq (266 µCi) [14C] (Treatment C) in the fed state following a standard breakfast on the morning of Day 1.

A subject in Part 2 will be considered evaluable if they had provided biological samples for up to 168 hours after drug administration or demonstrates >90% mass balance recovery, or < 1% of the administered dose eliminated in excreta for 2 consecutive days, whichever was sooner.

Approximately 7 days after subjects are discharged from Part 1 of the study, subjects are to be admitted to the clinical unit on the evening of the day prior to IMP administration (Day -1 of Part 2) for confirmation of eligibility and baseline procedures.

Subjects are to be dosed on the morning following admission (Day 1 of Part 2). Following an overnight fast (approximately 10 h), subjects consume a standard breakfast and receive a single dose of [14C]-KD025 200 mg Capsule (Treatment C) 30 min after the start of breakfast. Subjects are to remain in the clinic until up to 168 hours after dosing (up to Day 8 of Part 2). The plan is for subjects to be released as a group when all subjects had achieved a mass balance cumulative recovery of > 90% or if < 1% of the dose administered had been collected in urine and feces within 2 separate consecutive 24-hour periods. This may result in the subjects being discharged as a group prior to completion of the planned residency period. Once the discharge criteria or the planned residency period is achieved, the subjects are to undergo discharge assessments; collection of all samples (blood, urine and feces) is stopped.

If mass balance criteria has not been met by all subjects on Day 8, the residency period for the subjects not achieving the release criteria may be extended up to a maximum of 216 h post-dose (Day 10 of Part 2). During the additional residency period, only urine and/or feces are to be collected. If the criterion is still not met by Day 10, or if additional residency not considered appropriate or necessary, then home collections of urine and/or feces may be requested at the discretion of the Investigator for individual subjects. To ensure ongoing well-being of subjects, a follow-up phone call will take place 5 to 7 days post-discharge from the study or after the end of the last collection period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination), electrocardiogram (ECG) and laboratory investigations (hematology, clinical chemistry and urinalysis)
3. Body weight ≥ 50 kg
4. Body mass index (BMI) of 18.0 to 35.0 kg/m^2
5. Must be willing and able to communicate and participate in the whole study
6. Must have regular bowel movements (i.e., average stool production of ≥ 1 and ≤ 3 stools per day)
7. Subjects must have participated in Part 1 in order to be eligible for Part 2
8. Must provide written informed consent
9. Must agree to adhere to the contraception requirements of the study

In addition to the above criteria, subjects must agree to the following restrictions:

* No alcohol during the 24 hours prior to screening and the 24-hour prior to each admission until discharge from each part of the study.
* No food or drinks containing grapefruit, cranberry, caffeine or other xanthines from 24 hours prior to each admission until discharge from each part of the study.
* No food containing poppy seeds for 48 hours prior to screening and for 48 hours prior to each admission until discharge from each part of the study.
* No unaccustomed strenuous exercise from the 72-hour period before the screening visit and then from 72 hours prior to each admission until discharge from each part of the study.

Exclusion Criteria:

1. Subjects who previously participated in any other investigational study drug trial in which receipt of an investigational study drug occurred within 90 days prior to dosing
2. Subjects who have previously participated in a study where subjects were dosed with belumosudil
3. Subjects who are study site employees or immediate family members of a study site or sponsor employee
4. Subjects with pregnant partners
5. History of any drug or alcohol abuse in the past 2 years
6. Regular alcohol consumption in males > 21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
7. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission
8. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
9. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionizing Radiation Regulations 2017.
10. Subjects who have been enrolled in an ADME/IV microtracer study in the last 12 months
11. Subjects who do not have suitable veins for multiple venepunctures/cannulation
12. Clinically significant abnormal biochemistry, hematology or urinalysis. Subjects with blood platelet count, hemoglobin and red blood cells lower than the reference range
13. Confirmed positive drugs of abuse test result
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV) results
15. Evidence of renal impairment at screening as indicated by an estimated creatinine clearance of < 80 mL/min using the Cockcroft-Gault equation
16. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal (GI) disease, neurological or psychiatric disorder, as judged by the Investigator
17. Subject has a history or presence of any of the following:

    * Active GI disease requiring therapy
    * Hepatic disease and/or alanine aminotransaminase or aspartate aminotransaminase > upper limit of normal (ULN)
    * Renal disease and/or serum creatinine > upper limit of normal (ULN)
    * Other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
18. Subject has QT interval corrected using Fridericia's formula (QTcF) intervals > 450 msec at screening or admission
19. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
20. Presence or history of clinically significant allergy requiring treatment
21. Donation or loss of greater than 400 mL of blood within the previous 3 months
22. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies in the 14 days before study drug administration.
23. Failure to satisfy the Investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy males
Enrollment: 5 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Ltd, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schueller O, Skucas E, Regev G, Shaw I, Singh N, Sanghvi M, Croft M, Lohmer L, Alabanza A, Patel J. Absolute Bioavailability, Mass Balance, and Metabolic Profiling Assessment of [14 C]-Belumosudil in Healthy Men: A Phase 1, Open-Label, 2-Part Study. Clin Pharmacol Drug Dev. 2022 Jul;11(7):786-794. doi: 10.1002/cpdd.1085. Epub 2022 Mar 1. PMID 35231159

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects (Part 1 and Part 2): Part 1: (Treatment A) KD025 200 mg tablet, fed (Day 1). then 1.75 hours later (Treatment B) [14C]-KD025 solution for infusion, 20 μg/mL (100 μg in 5 mL), containing not more than 37 kBq (1000 nCi) [14C], as a 15 min IV infusion, 100 μg, fed
  Part 2: (Treatment C) Single [14C]-KD025 capsule 200 mg containing <= 9.8 megabecquerel 14C, fed
Period: Overall Study
Arm/Group | All Subjects (Part 1 and Part 2)
Started | 5
Completed Part 1 | 5
Completed Part 2 | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects who received a single dose [14C]-KD025 and oral belumosudil tablet
Arm/Group | All Subjects
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.86 (3.06)

OUTCOME MEASURES:

1. Primary Outcome: Part 1 Pharmacokinetics: t(1/2) for Belumosudil Tablet and [14C]-KD025 IV
Description: Apparent terminal elimination half-life (t[1/2] for Part 1: (Treatment A) KD025 200 mg tablet, fed (Day 1). then 1.75 hours later (Treatment B) [14C]-KD025 solution for infusion 20 microgm/mL (100 microgm in 5 mL) containing <= 37 kilobecquerel as 15 min IV infusion 100 microgm, fed
Time Frame: Plasma samples belumosudil relative to oral dosing: 0,0.5,1,1.5,2,3,4,5,6,8,10,12,24,36, and 48 hours post-dosing. Plasma samples [14C]-KD025 relative to end infusion:-0.25,-0.16,-0.08,0,0.08,0.16,0.25,0.5,0.75,1,1.5,2,3,4,5,6,8,10,12,22,34, and 46 h
Population: All subjects
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Groups:
- Part 1: Treatment A: Belumosudil 200 mg Tablet
- Part 1: Treatment B: [14C]-KD025 at a dose of 100 μg in a 5 mL solution IV (20 μg per mL)
Arm/Group | Part 1: Treatment A | Part 1: Treatment B
Number analyzed (Participants) | 5 | 5
Hours | 5.298 (66.7) | 5.857 (35.8)

2. Secondary Outcome: Part 1 Pharmacokinetics: Tmax for Belumosudil Tablet and [14C]-KD025
Description: Part 1: Time of maximum plasma concentration (Tmax) for belumosudil 200 mg oral tablet and [14C]-KD025 at a dose of 100 μg in a 5 mL solution IV
Time Frame: Plasma samples belumosudil relative oral dosing: 0,0.5,1,1.5,2,3,4,5,6,7,8,10,12,24,36, and 48 hours post-dosing. Plasma samples [14C]-KD025 relative to end infusion:-0.25,-0.16,-0.08,0,0.08,0.16,0.25,0.5,0.75,1, 1.5,2,3,4,5,6,8,10,12,22,34,and 46 h
Measure: Median (Full Range); unit: Hours
Groups:
- Part 1: Treatment B: [14C]-KD025 at a dose of 100 μg in a 5 mL solution IV
Arm/Group | Part 1: Treatment A | Part 1: Treatment B
Number analyzed (Participants) | 5 | 5
Hours | 2.000 [1.00 to 4.00] | 0.248 [0.24 to 0.25]

3. Secondary Outcome: Part 1 Pharmacokinetics: Cmax of Belumosudil Tablets
Description: The maximum concentration (Cmax) of belumosudil 200 mg tablets
Time Frame: Plasma samples belumosudil relative to oral dosing: 0,0.5,1,1.5,2,3,4,5,6,7,8,10,12,24,36, and 48 hours post-dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1 Treatment A: Belumosudil 200 mg Tablet 200 mg
Arm/Group | Part 1 Treatment A
Number analyzed (Participants) | 5
ng/mL | 1870 (36.7)

4. Secondary Outcome: Part 1 Pharmacokinetics: Cmax of [14C]-KD025 IV
Description: The maximum concentration (Cmax) of belumosudil [14C]-KD025 at a dose of 100 μg in a 5 mL solution IV
Time Frame: Plasma samples for [14C]-KD025 relative to end of infusion:-0.25,-0.16,-0.08,0,0.08,0.16,0.25,0.5,0.75,1, 1.5,2,3,4,5,6,8,10,12,22,34,46 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pg/mL)/(ng equiv/mL)
Arm/Group | Part 1: Treatment B
Number analyzed (Participants) | 5
(pg/mL)/(ng equiv/mL) | 4480 (18.0)

5. Secondary Outcome: Part 1 Pharmacokinetics: AUC(0-inf) of Belumosudil Tablets
Description: The area under the concentration-time curve from zero extrapolated to infinity (AUC[0-inf]) of belumosudil 200 mg tablets
Time Frame: Plasma samples for belumosudil relative to oral dosing: 0,0.5,1,1.5,2,3,4,5,6,7,8,10,12,24,36, and 48 hours post-dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h)/mL
Groups:
- Part 1 Treatment A: Belumosudil 200 mg Tablet, 200 mg
Arm/Group | Part 1 Treatment A
Number analyzed (Participants) | 5
(ng*h)/mL | 8300 (40.2)

6. Secondary Outcome: Part 1 Pharmacokinetics: AUC(0-inf) of [14C]-KD025 IV
Description: The area under the concentration-time curve from zero extrapolated to infinity (AUC[0-inf]) of [14C]-KD025 at a dose of 100 μg in a 5 mL solution IV
Time Frame: Plasma samples for [14C]-KD025 relative to end of infusion:-0.25,-0.16,-0.08,0,0.08,0.16,0.25,0.5,0.75,1, 1.5,2,3,4,5,6,8,10,12,22,34,and 46 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ((ng*h)/mL)/(ng equiv*h/mL)
Arm/Group | Part 1: Treatment B
Number analyzed (Participants) | 5
((ng*h)/mL)/(ng equiv*h/mL) | 6480 (29.3)

7. Secondary Outcome: Part 1: Absolute Bioavailability of Belumosudil 200 mg Tablet
Description: The absolute bioavailability following oral administration of belumosudil 200 mg tablet, based on the area under the concentration-time curve from zero dosing extrapolated to infinity (AUC[0-inf])
Time Frame: Plasma samples for belumosudil relative to oral dosing: 0,0.5,1,1.5,2,3,4,5,6,7,8,10,12,24,36, and 48 hours post-dosing.
Measure: Number; unit: Percentage
Arm/Group | Part 1: Treatment A
Number analyzed (Participants) | 5
Percentage | 64

8. Secondary Outcome: Part 2: Mass Balance Recovery Following 200 mg Oral Dose of [14C]-KD025 Capsule
Description: Cumulative amount of total radioactivity excreted and recovered in urine, feces and total excreta (urine and feces combined) following dosing with [14C]-KD025 200 mg oral capsule.
Time Frame: Cumulative sample collection time frame 0-6 hours, 0-12 hours, 0-24 hours, 0-48 hours, 0-72 hours, 0-96 hours, 0-120 hours, 0-144 hours, 0-168 hours, 0-192 hours, 0-216 hours post-dose
Measure: Number; unit: Percentage
Groups:
- Cumulative Urine Ae(%): Percentage of [14C]-KD025 200 mg oral capsule excreted in urine
- Cumulative Feces Ae (%): Percentage of [14C]-KD025 200 mg oral capsule excreted in feces
- Cumulative Total Ae (%): Percentage of [14C]-KD025 200 mg oral capsule excreted overall
Arm/Group | Cumulative Urine Ae(%) | Cumulative Feces Ae (%) | Cumulative Total Ae (%)
Number analyzed (Participants) | 5 | 5 | 5
Percentage
  0-6 (hours) | 2.194 | NA — Feces sample only collected once per day and reported in the 0-24 hour period. | NA — Feces sample only collected once per day and reported in the 0-24 hour period.
  0-12 (hours) | 3.343 | NA — Feces sample only collected once per day and reported in the 0-24 hour period. | NA — Feces sample only collected once per day and reported in the 0-24 hour period.
  0-24 (hours) | 3.773 | 27.431 | 31.203
  0-48 (hours) | 3.933 | 75.499 | 79.432
  0-72 (hours) | 3.958 | 81.597 | 85.555
  0-96 (hours) | 3.966 | 83.044 | 87.010
  0-120 (hours) | 3.972 | 84.070 | 88.042
  0-144 (hours) | 3.976 | 84.340 | 88.315
  0-168 (hours) | 3.977 | 84.436 | 88.413
  0-192 (hours) | 3.979 | 84.493 | 84.472
  0-216 (hours) | 3.980 | 84.553 | 88.533

9. Secondary Outcome: Part 2 Pharmacokinetics: Tmax of 200 mg [14C]-KD025
Description: Time of maximum concentration (Tmax) following a single oral dose of 200 mg [14C]-KD025 capsule
Time Frame: Time Relative to Belumosudil Dosing: 0,0.5,1,1.5,2,3,4,5,6,8,10,12,24,36,48,72,96,120,144, and 168 hours post-dose
Measure: Median (Full Range); unit: Hours
Groups:
- [14C]-KD025 Oral 200 mg KD025: [14C]-KD025 200 mg belumosudil oral capsule in the fed state
Arm/Group | [14C]-KD025 Oral 200 mg KD025
Number analyzed (Participants) | 5
Hours | 2.000 [1.50 to 2.05]

10. Secondary Outcome: Part 2 Pharmacokinetics: t(1/2) of 200 mg [14C]-KD025
Description: Apparent terminal elimination half-life (t[1/2]) following a single oral dose of 200 mg [14C]-KD025 capsule
Time Frame: Time Relative to Belumosudil Dosing: 0,0.5,1,1.5,2,3,4,5,6,8,10,12,24,36,48,72,96,120,144, and 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-KD025 Oral 200 mg KD025
Number analyzed (Participants) | 5
Hours | 5.109 (37.9)

11. Secondary Outcome: Part 2 Pharmacokinetics: Cmax of 200 mg [14C]-KD025
Description: Maximum concentration following a single oral dose of 200 mg [14C]-KD025 capsule
Time Frame: Time Relative to Belumosudil Dosing: 0,0.5,1,1.5,2,3,4,5,6,8,10,12,24,36,48,72,96,120,144, and 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-KD025 Oral 200 mg KD025
Number analyzed (Participants) | 5
ng/mL | 1680 (32.1)

12. Secondary Outcome: Part 2 Pharmacokinetics: AUC(0-inf) of 200 mg [14C]-KD025
Description: Area under the concentration-time curve from zero dosing extrapolated to infinity following a single oral dose of 200 mg [14C]-KD025 capsule
Time Frame: Time Relative to Belumosudil Dosing: 0,0.5,1,1.5,2,3,4,5,6,8,10,12,24,36,48,72,96,120,144, and 168 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h)/mL
Arm/Group | [14C]-KD025 Oral 200 mg KD025
Number analyzed (Participants) | 5
(ng*h)/mL | 8100 (37.0)

ADVERSE EVENTS:
Time Frame: Up to 20 days
Groups:
- All Subjects: All subjects completing Part 1 and Part 2
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results. The sponsor cannot require changes to the study results in the communication except to remove sponsor's confidential information. Sponsor cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT03907540/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03907540/SAP_001.pdf